CLINICAL TRIAL: NCT05772143
Title: Percutaneous Lumbar Discectomy : Evaluation of Patient Reported Outcomes, Aconomical Impact and Return to Work
Brief Title: Percutaneous Discectomy to Treat Symptomatic Lumbar Disc Herniation : Evaluation of Clinical Efficiency, Patient Reported Outcomes and Economical Impact by Assessing Time Before Return to Work and Duration of Hospitalization Stay
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Imagerie01
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lumbar disc herniation: Patient over 18 years of age suffering from radiculalgia related to lumbar disc herniation visualized on MRI with radio-clinical concordance, failure of conservative treatment and nerve root infiltrations
  Interventions: Procedure: Percutaneous discectomies under CT

INTERVENTIONS:
Procedure: Percutaneous discectomies under CT — Percutaneous discectomies under CT guidance to treat lumbar disc herniations resistant to conservative treatment and nerve root infiltrations.

SUMMARY:
This study aims to evaluate the clinical (pain) and functional (patient reported outcomes) efficacy of percutaneous discectomies under CT guidance to treat lumbar disc herniations resistant to conservative treatment and nerve root infiltrations.

The aim is also to evaluate the economic impact of the procedure, mainly through the length of hospitalization and the time to return to work.

Patients were evaluated initially before surgery and then at 1, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* radiculalgia related to lumbar disc herniation with clinical radiological concordance
* age > 18
* resistance to conservative treatment and nerve root infiltrations

Exclusion Criteria:

* prior discal surgery at the same level,
* lumbar canal stenosis,
* extruded discal herniation,
* neurological deficit,
* no capacity to answer to follow-up calls

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years of age suffering from radiculalgia related to lumbar disc herniation visualized on MRI with radio-clinical concordance, failure of conservative treatment and nerve root infiltrations ; consulting in interventionnal radiology care unit,
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index | before treatment
  Fonctionnal indicator of incapicity validated for patient suffering from spinal disorders
Oswestry disability index | At 1 month after treatment
  Fonctionnal indicator of incapicity validated for patient suffering from spinal disorders
Oswestry disability index | At 3 month after treatment
  Fonctionnal indicator of incapicity validated for patient suffering from spinal disorders
Oswestry disability index | At 6 month after treatment
  Fonctionnal indicator of incapicity validated for patient suffering from spinal disorders

SECONDARY OUTCOMES:
Visual analogic scale | Initially and at 1 month, 3 month and 6 month after the procedure
  pain rating scale from 0 to 10 (worst is 10)
Off work duration | Initially and at 1 month, 3 month and 6 month after the procedure
  days before returning to work
Hospitalization duration | Initially and at 1 month, 3 month and 6 month after the procedure
  overnights hospitalization stays following the intervention
use of pain killers | Initially and at 1 month, 3 month and 6 month after the procedure
  frequency of the use of painkillers before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No
Not scheduled

REFERENCES:
- [Derived] Ranc PA, Rudel A, Bentellis I, Prestat A, Elbaze S, Sala V, Torre F, Pavan LJ, Uri IF, Amoretti N. Patient-Reported Outcomes and Return to Work after CT-Guided Percutaneous Lumbar Discectomy: A Prospective Study. J Vasc Interv Radiol. 2024 Mar;35(3):390-397. doi: 10.1016/j.jvir.2023.12.007. Epub 2023 Dec 16. PMID 38110149